CLINICAL TRIAL: NCT07040098
Title: A Prospective, Multicenter, Randomized Clinical Trial of Optimizing Immunotherapy Combined With Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer (STELLARIII)
Brief Title: Optimizing Immunotherapy Combined With Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer
Acronym: STELLARIII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, JIN JING, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5362
Record Dates: First submitted 2025-05-20; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: Locally advanced rectal cancer; TNT; Immunotherapy; CR rate
MeSH Terms: interventions — sintilimab; Immune Checkpoint Inhibitors; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group SCRT-4 (Experimental): The intervention of group SCRT-4 is Short-course radiotherapy followed by neoadjuvant chemotherapy and PD-1 inhibitor, which consists of a short-course radiotherapy(SCRT, 5 Gy x 5 alone), then after 14 days of radiotherapy completed, four cycles of PD-1 inhibitor and four cycles of CAPOX will be performed. The regimen of PD-1 inhibitor and CAPOX treatment includes Sintilimab 200 mg IV, day 1，Oxaliplatin 130 mg/m2 IV day 1，Capecitabine 1000 mg/m2 twice daily PO for 14 days(3 weeks per cycle).Then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Drug: Sintilimab; Radiation: Short-course radiotherapy; Combination Product: CAPOX
- Group SCRT-6 (Experimental): The intervention of group SCRT-6 is Short-course radiotherapy followed by neoadjuvant chemotherapy and PD-1 inhibitor, which consists of a short-course radiotherapy(SCRT, 5 Gy x 5 alone), then after 14 days of radiotherapy completed, six cycles of PD-1 inhibitor and six cycles of CAPOX will be performed. The regimen of PD-1 inhibitor and CAPOX treatment includes Sintilimab 200 mg IV, day 1，Oxaliplatin 130 mg/m2 IV day 1，Capecitabine 1000 mg/m2 twice daily PO for 14 days(3 weeks per cycle).Then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Drug: Sintilimab; Radiation: Short-course radiotherapy; Combination Product: CAPOX
- Group LCRT-4 (Experimental): The intervention of group LCRT-4 is Long-course concurrent chemoradiotherapy followed by neoadjuvant chemotherapy and PD-1 inhibitor, which consists of a Long-course concurrent chemoradiotherapy (LCRT, 2 Gy x 25f, concurrently with capecitabine 825 mg/m2, twice a day), then after 14 days of radiotherapy completed, four cycles of PD-1 inhibitor and four cycles of CAPOX will be performed. The regimen of PD-1 inhibitor and CAPOX treatment includes Sintilimab 200 mg IV, day 1，Oxaliplatin 130 mg/m2 IV day 1，Capecitabine 1000 mg/m2 twice daily PO for 14 days(3 weeks per cycle).Then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Drug: Sintilimab; Radiation: Long-course concurrent chemoradiotherapy; Combination Product: CAPOX
- Group LCRT-6 (Experimental): The intervention of group LCRT-6 is Long-course concurrent chemoradiotherapy followed by neoadjuvant chemotherapy and PD-1 inhibitor, which consists of a Long-course concurrent chemoradiotherapy (LCRT, 2 Gy x 25f, concurrently with capecitabine 825 mg/m2, twice a day), then after 14 days of radiotherapy completed, six cycles of PD-1 inhibitor and six cycles of CAPOX will be performed. The regimen of PD-1 inhibitor and CAPOX treatment includes Sintilimab 200 mg IV, day 1，Oxaliplatin 130 mg/m2 IV day 1，Capecitabine 1000 mg/m2 twice daily PO for 14 days(3 weeks per cycle).Then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Drug: Sintilimab; Radiation: Long-course concurrent chemoradiotherapy; Combination Product: CAPOX

INTERVENTIONS:
Drug: Sintilimab — PD-1 inhibitor
  Other Names: Immune checkpoint inhibitor
Radiation: Short-course radiotherapy — Pelvic radiation, SCRT, 5 Gy x 5 alone
  Other Names: hypofraction
  Arms: Group SCRT-4; Group SCRT-6
Radiation: Long-course concurrent chemoradiotherapy — Pelvic radiation, 50 Gy in 25 fractions over 5 weeks, concurrently with capecitabine (825 mg/m2, twice a day).
  Other Names: CCRT
  Arms: Group LCRT-4; Group LCRT-6
Combination Product: CAPOX — chemotherapy regimen, Oxaliplatin 130 mg/m2 IV day 1，Capecitabine 1000 mg/m2 twice daily PO for 14 days(3 weeks per cycle)
  Other Names: neoadjuvant chemotherapy

SUMMARY:
This study explores the key clinical issues in the field of neoadjuvant therapy for locally advanced rectal cancer. There are three core problems with the currently recommended total neoadjuvant therapy (TNT) in the guidelines: the lack of evidence-based consensus on the timing of radiotherapy and chemotherapy, the undefined number of chemotherapy cycles, and the uncertainty in the selection of the precise radiotherapy mode. In recent years, the combination of immune checkpoint inhibitors (ICIs) with the PD-1/PD-L1 inhibitors as the core and the TNT regimen has shown a trend of further enhancing tumor regression, providing a possibility for the organ function preservation of rectal cancer. However, existing clinical studies exhibit a high degree of heterogeneity in treatment strategies. In particular, there is a lack of high-quality evidence-based medical evidence in core aspects such as the timing of ICIs intervention and the combination of treatment regimens. This study is designed as a prospective, multicenter, randomized controlled phase II study. The "pick the winner" strategy for screening the optimal regimen is adopted to evaluate the efficacy of four neoadjuvant regimens (Group SCRT-4: short-course radiotherapy → 4 cycles of chemotherapy + ICIs; Group SCRT-6: short-course radiotherapy → 6 cycles of chemotherapy + ICIs; Group LCRT-4: concurrent chemoradiotherapy → 4 cycles of chemotherapy + ICIs; Group LCRT-6: concurrent chemoradiotherapy → 6 cycles of chemotherapy + ICIs). By evaluating indicators such as the complete response rate, organ preservation rate, safety, long-term survival, as well as the anal function and quality of life of patients, treatment strategies with clinical advantages will be screened out, providing an evidence-based basis for subsequent phase III confirmatory trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, regardless of gender;
2. Pathologically confirmed rectal adenocarcinoma with immunohistochemical results indicating pMMR (proficient mismatch repair) or genetic testing confirming MSS (microsatellite stability);
3. Staged as clinical stage II/III (cT3-T4N0 or cT2-4N+, no distant metastasis, per the 8th Edition AJCC Cancer Staging Manual, 2018) via MRI or endoscopic ultrasound, and meeting any one of the following:

   * cT3 with tumor inferior margin ≤ 6 cm from the anal verge;

     * cT3c/d with tumor inferior margin ≥ 6-12 cm from the anal verge; ③ cN2; ④ cT4; ⑤ MRF+ (mesorectal fascia involvement); ⑥ EMVI+ (extramural vascular invasion);
4. ECOG performance status 0-1;
5. Meeting basic laboratory criteria (e.g., hematologic, hepatic, and renal function);
6. No history of hypersensitivity to 5-Fu-based agents or platinum-based drugs;
7. Patients with primary rectal cancer must have received no prior surgery (excluding palliative colostomy), chemotherapy, or other antitumor therapies from diagnosis to enrollment;
8. No prior radiation to the planned radiotherapy site;
9. Signed informed consent form.

Exclusion Criteria:

1. Prior treatment with anti-PD-1/L1 and/or anti-CTLA-4 immunotherapy or other investigational immunotherapeutic agents;
2. History of severe autoimmune diseases, including active inflammatory bowel disease (IBD) (e.g., Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (e.g., granulomatosis with polyangiitis);
3. Symptomatic interstitial lung disease or active infectious/non-infectious pneumonitis;
4. Risk factors for bowel perforation, such as active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis, or other known predisposing conditions;
5. History of other malignancies, except for cured non-melanoma skin cancer or cervical carcinoma in situ;
6. Active infection, heart failure, myocardial infarction within 6 months, unstable angina, or uncontrolled arrhythmia;
7. Physical examination findings or clinical laboratory abnormalities deemed by the investigator to interfere with study outcomes or increase treatment-related risks, or other uncontrolled comorbidities;
8. Pregnant or breastfeeding women;
9. Congenital or acquired immunodeficiency disorders, including HIV infection, or history of organ/stem cell transplantation;
10. Active hepatitis B (HBV-DNA ≥2000 U/mL), hepatitis C (HCV), or active tuberculosis infection;
11. Prior administration of cancer vaccines or receipt of any vaccine within 4 weeks before treatment initiation (Note: Seasonal inactivated influenza vaccines are permitted; live-attenuated intranasal vaccines are prohibited);
12. Concurrent use of immunomodulators, chemotherapy, investigational drugs, or long-term corticosteroids (≥10 mg/day prednisone equivalent);
13. Patients with psychiatric disorders, substance abuse, or social circumstances that may compromise compliance, as assessed by the investigator;
14. Hypersensitivity or contraindications to the study medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete response | 2 months after completion of neoadjuvant therapy or 10 days after surgery
  The rate of pathological complete response plus clinical complete response

SECONDARY OUTCOMES:
Rate of TRG grade | 10 days after surgery
  Dowrak TRG grade
Tumor downstaging rate | 10 days after surgery
  rate of ypT0-2N0
Rate of acute toxicities during radiation, chemotherapy ± immunotherapy | 1 week after completion of neoadjuvant therapy
  Incidence of acute toxicities during radiation, chemotherapy ± immunotherapy
Rate of surgical complications | 3 months after completion of surgery
  Clavien-Dindo Grade
Rate of OS | 3 years after randomization
  overall survival
Rate of DFS | 3 years after randomization
  Disease-Free Survival
Rate of LRR | 3 years after randomization
  Locoregional Recurrence
Rate of DM | 3 years after randomization
  Distant Metastasis
Organ Preservation Rate | 3 years after randomization
  The organ preservation rate is defined as the proportion of patients who successfully retain the rectal organ and its function through effective local treatment of the primary lesion, achieved by approaches such as a watch-and-wait (W&W) strategy or local excision. Successful organ preservation is determined if the following criteria are met:
  1. Undergoing the W&W approach without local regrowth;
  2. Undergoing local excision with negative resection margins and no local recurrence;
  3. Avoidance of total mesorectal excision (TME) surgery with preservation of functional rectal reflex pathways;
  4. No definitive evidence of residual local tumor;
  5. Absence of a permanent stoma or unclosed temporary stoma.
Quality of life (QoL) in cancer patients | baseline, 10 days after completion of neoadjuvant therapy, 10 days after surgery, 3 months after randomization, 6 months after randomization, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Quality of life in cancer patients will be evaluated using the European Organisation for Treatment and Research of Cancer (EORTC) Quality of Life Questionnaires QLQ-C30 . The scoring and interpretation of the QLQ-C30 scales were performed according to the EORTC guidelines. Each item is scored from 0 to 100, with higher scores indicating better functioning on the functional scales/items and more severe symptoms on the symptom scales/items.
Quality of life (QoL) in rectal cancer patients | baseline, 10 days after completion of neoadjuvant therapy, 10 days after surgery, 3 months after randomization, 6 months after randomization, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Quality of life in rectal cancer patients will be evaluated using the European Organisation for Treatment and Research of Cancer (EORTC) Quality of Life Questionnaires QLQ-CR29 . The scoring and interpretation of the QLQ-CR29 scales were performed according to the EORTC guidelines. Each item is scored from 0 to 100, with higher scores indicating better functioning on the functional scales/items and more severe symptoms on the symptom scales/items.
Anal function | baseline, 10 days after completion of neoadjuvant therapy, 10 days after surgery, 3 months after randomization, 6 months after randomization, 1 year after randomization, 2 years after randomization, 3 years after randomization
  Anal function will be evaluated using the Wexner incontinence score. This scoring system consists of 5 items evaluating the frequency of gas incontinence, frequency of liquid incontinence, frequency of solid incontinence, frequency of wearing pads, and lifestyle alterations, with a score ranging from 0-4 for each question. The total score is calculated, with higher scores indicating poorer anal function.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing
  - National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital & Shenzhen Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: No